CLINICAL TRIAL: NCT02271035
Title: A Prospective Study Comparing the Success Rate of Injection of Dextranomer /Hyaluronic Acid (DefluxR) Versus Polyacrylate Polyalcohol (VantrisR) for Treatment of Bilateral Similar Grade Vesicoureteral Reflux in Children
Brief Title: A Prospective Study Comparing the Success Rate of Injection of (DefluxR) Versus (VantrisR) for VUR in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Rabin Medical Center
Record Dates: First submitted 2013-08-15; First posted 2014-10-22 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-06

CONDITIONS: Vesico-Ureteral Reflux
Keywords: VUR
MeSH Terms: conditions — Vesico-Ureteral Reflux | interventions — deflux; dextranomer; Hyaluronic Acid; Vantris; polyacrylate polyalcohol copolymer

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Deflux (Active Comparator): In each patient, Deflux will be injected into one of the ureteral orifices using the the HIT technique.
  Interventions: Drug: Deflux
- Vantris (Active Comparator): Vantris will be injected into the other ureteral orifice using the same technique and the same amount of implant.
  Interventions: Drug: Vantris

INTERVENTIONS:
Drug: Deflux — Deflux will be injected through the working channel of the cystoscope using a special needle into the submucosal space of the ureteral orifice (Deflux to one ureteral orifice and Vantris to the other side). The technique that will be used is HIT (Hydrodistention Implantation Technique)+ STING
  Other Names: Dextranomer/hyaluronic acid
  Arms: Deflux
Drug: Vantris — vantris will be injected through the working channel of the cystoscope using a special needle into the submucosal space of the ureteral orifice (Deflux to one Vantris to the other side). The technique that will be used is HIT (Hydrodistention Implantation Technique)+ STING
  Other Names: Polyacrylate Polyalcohol copolymer
  Arms: Vantris

SUMMARY:
Vesicoureteral reflux (VUR) is the most common urologic diagnosis in neonates estimated at 1% of newborns, and 30-45% of the children who present with urinary tract infection (1).

Optional treatments of children with VUR include conservative therapy with or without prophylactic antibiotics, and endoscopic, laparoscopic, or open surgery.

In an endoscopic technique, the injecting needle is inserted through the working channel of the cystoscope. The procedure is relatively short and is performed as out-patient surgery.

In 2000, Dextranomer/Hyaluronic acid (DefluxR) was approved by the FDA, and subsequently has become the treatment of choice in VUR grades 2-4.

In 2004, the hydrodistention-implantation technique (HIT) was introduced by Kirsch. HIT involves the use of a pressurized stream of fluid directed into the ureter to aid visualization, and injection into the submucosa within the ureteric tunnel to improve coaptation of the ureter (3).

One of the disadvantages attributed to Deflux is the loss of 20% of the injected material over time (a result of absorption of the hyaluronic acid), which may explain the lower success rate of the endoscopic treatment of VUR compared with open surgery.

In 2005, Polyacrylate Polyalcohol (VantrisR), a non- absorbable chemical preparation was introduced for endoscopic treatment of VUR, aiming to improve on the results of Deflux by preventing volume loss. Preliminary results of a three year follow-up using Vantris have shown high a level of reflux resolution(4).

The aim of the current study is to compare the rate of resolution of the VUR using Deflux versus Vantris in bilateral VUR

DETAILED DESCRIPTION:
Vesicoureteral reflux (VUR) is the most common urologic diagnosis in neonates estimated at 1% of newborns, and 30-45% of the children who present with urinary tract infection (1).

Optional treatments of children with VUR include conservative therapy with or without prophylactic antibiotics, and endoscopic, laparoscopic, or open surgery.

The first endoscopic treatment was presented in 1981 by Matouschek, who injected Teflon into the submucosa of the ureteral orifice, at the six o'clock position (STING). In this technique, the injecting needle is inserted through the working channel of the cystoscope. The procedure is relatively short and is performed as out-patient surgery.

In 2000, Dextranomer/Hyaluronic acid (DefluxR) was approved by the FDA, and subsequently has become the treatment of choice in VUR grades 2-4.

In 2004, the hydrodistention-implantation technique (HIT) was introduced by Kirsch. HIT involves the use of a pressurized stream of fluid directed into the ureter to aid visualization, and injection into the submucosa within the ureteric tunnel to improve coaptation of the ureter (3).

A review of Deflux therapy for VUR in 63 studies, including 8101 ureters, found a success rate of 51%-79% depending on VUR grade. (grade 1,2 79%, grade 3 72%, grade 4 63%, grade 5 51%) (2).

One of the disadvantages attributed to Deflux is the loss of 20% of the injected material over time (a result of absorption of the hyaluronic acid), which may explain the lower success rate of the endoscopic treatment of VUR compared with open surgery.

In 2005, Polyacrylate Polyalcohol (VantrisR), a non- absorbable chemical preparation was introduced for endoscopic treatment of VUR, aiming to improve on the results of Deflux by preventing volume loss. Preliminary results of a three year follow-up using Vantris have shown high a level of reflux resolution(4).

The aim of the current study is to compare the rate of resolution of the VUR using Deflux versus Vantris in bilateral VUR

ELIGIBILITY:
Inclusion Criteria:

* Bilateral VUR of the same grade

Exclusion Criteria:

* Inability to apply the same technique on both ureteral orifices

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
rate of resolution of VUR using Vantris vs.Deflux | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David Ben-Meir, MD, Principal Investigator — Investigator
Locations (1):
- Schneider Medical Center of Israel, Petah Tikva, Israel, Israel